CLINICAL TRIAL: NCT03564262
Title: Effects of Acute Dietary Sodium on Cerebrovascular Reactivity and Blood Pressure Reactivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, William Farquhar, Professor, University of Delaware
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 1178955-1
Record Dates: First submitted 2018-05-16; First posted 2018-06-20 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Blood Pressure; Cerebrovascular Reactivity
MeSH Terms: interventions — Sodium

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cerebrovascular Reactivity (Experimental): Cerebrovascular reactivity (CVR) will be assessed using transcranial Doppler ultrasound with carbon dioxide as the vasoactive stimuli.
  The intervention is to provide subjects with either a low sodium meal (138 mg sodium) and high sodium meal (1,495 mg sodium), in a randomized order. The CVR test will be performed prior to soup consumption as well as after soup consumption.
  Interventions: Other: Low Sodium Meal (138 mg sodium); Other: High Sodium Meal (1,495 mg sodium)
- Blood Pressure Reactivity (Experimental): Blood pressure responses during dynamic exercise will be assessed. The intervention is to provide subjects with either a low sodium meal (138 mg sodium) and high sodium meal (1,495 mg sodium), in a randomized order. Blood pressure reactivity during dynamic exercise will be assessed after soup consumption.
  Interventions: Other: Low Sodium Meal (138 mg sodium); Other: High Sodium Meal (1,495 mg sodium)

INTERVENTIONS:
Other: Low Sodium Meal (138 mg sodium) — One Low Sodium Meal
Other: High Sodium Meal (1,495 mg sodium) — One High Sodium Meal

SUMMARY:
Americans eat more salt than is recommended by the American Heart Association. This is important because consuming a high-salt diet is associated with an increased risk of cardiovascular events, like strokes and heart attacks. In fact, consuming one high-salt meal temporarily reduces blood vessel function and it is not uncommon for Americans to consume high-salt meals. Therefore, our laboratory is interested in determining if a single high-salt meal affects 1) brain blood vessel function at rest and 2) blood pressure responses during exercise.

DETAILED DESCRIPTION:
Excess dietary salt increases the risk of cardiovascular events like strokes and heart attacks, independent of resting blood pressure. Recent data found that consuming one high-salt meal temporarily reduces endothelial function in the periphery. This decrease in endothelial function can lead to an exaggerated blood pressure response during exercise and may also attenuate cerebrovascular reactivity at rest. This is essential, because an exaggerated cardiovascular response to exercise and a decrease in brain blood vessel function at rest are risk factors for future cardiovascular events. The long-term goal is to determine how dietary salt adversely affects BP and cerebrovascular regulation. The objective of this proposal is to evaluate the impact of an acute dietary salt meal on BP response during exercise and cerebrovascular reactivity at rest. The investigators have 2 specific aims: 1) Aim 1 will test the hypothesis that high dietary salt will reduce cerebrovascular reactivity, 2) Aim 2 will test the hypothesis that high dietary salt will augment blood pressure reactivity during exercise. The findings of this project will shed light on how acute dietary salt affects the risk of cardiovascular events during a bout of exercise and long-term risk for cardiovascular disease and stroke.

ELIGIBILITY:
Inclusion Criteria:

* normal blood pressure
* males, females, minorities

Exclusion Criteria:

* high blood pressure
* body mass index (BMI > 30 kg/m2)
* smokers or nicotine users
* those who are pregnant or planning to become pregnant
* allergy to the tomato soup

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Cerebrovascular Reactivity post soup consumption | Prior to and 60 minutes after soup consumption
  Middle Cerebral Artery/ End-tidal Carbon Dioxide (cm/s/mmHg)
Blood Pressure Reactivity- Dynamic Exercise | 80 minutes after soup consumption
  Change in Blood Pressure during dynamic exercise (mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: William B Farquhar, PhD, Principal Investigator — University of Delaware; Kamila U Migdal, BS, Principal Investigator — University of Delaware
Locations (1):
- William B Farquhar, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Migdal KU, Robinson AT, Watso JC, Babcock MC, Serrador JM, Farquhar WB. A high-salt meal does not augment blood pressure responses during maximal exercise. Appl Physiol Nutr Metab. 2020 Feb;45(2):123-128. doi: 10.1139/apnm-2019-0217. Epub 2019 Jun 25. PMID 31238011